CLINICAL TRIAL: NCT03189641
Title: An Exploratory Clinical Trial of Cilostazol Eluting Stent System (CES-1) in De Novo Coronary Artery Lesions
Brief Title: Clinical Trial of Cilostazol Eluting Stent System (CES-1) in De Novo Coronary Artery Lesions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: JIMRO Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JD-001
Record Dates: First submitted 2017-06-13; First posted 2017-06-16 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Coronary Artery Disease
Keywords: Drug eluting stents; Coronary artery disease; Coronary artery stenosis; Myocardial ischemia; Angioplasty
MeSH Terms: conditions — Coronary Artery Disease; Coronary Stenosis; Myocardial Ischemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Cilostazol eluting stent system (CES-1) (Experimental)
  Interventions: Device: Cilostazol eluting stent system (CES-1)

INTERVENTIONS:
Device: Cilostazol eluting stent system (CES-1) — Implantation of drug eluting stent

SUMMARY:
The purpose of the this trial is to evaluate the clinical safety and efficacy of Cilostazol eluting stent system (CES-1) for the treatment of single de novo lesions in native coronary arteries.

ELIGIBILITY:
Inclusion Criteria:

<Clinical selection criteria>

1. Patients who have provided written informed consent.
2. Patients who have evidence of myocardial ischemia confirmed by subjective symptoms (chest pain etc.), ST change in the electrocardiogram or objective findings.
3. Patients who are at least 20 years old.

<Angiographic selection criteria>

1. Single de novo lesion in native coronary arteries
2. Target vessel diameter is 2.75 mm to 3.25 mm.
3. TIMI flow is 2 or more.
4. Angiographic percent diameter stenosis (by visual estimation) is 75% or more in AHA classification

Exclusion Criteria:

<Clinical exclusion criteria>

1. Acute myocardial infarction Patients whose CK-MB or troponin exceeds the facility reference upper limit and have at least one of the following is confirmed are excluded as acute myocardial infarction.

   * Ischemic symptoms and Electrocardiographic findings showing continuous ischemia (eg, ST segment elevation or depression above 1 mm in contiguous leads, or the appearance of a new left bundle branch block).
   * Pathological Q waves on electrocardiogram
   * Myocardial necrotic focus or wall motion abnormality newly confirmed in diagnostic imaging
2. Patients who cannot be given emergency coronary artery bypass grafting (CABG).
3. Patients who cannot be administered antiplatelet drugs. The following cases are conceivable.

   * Significant intracranial hemorrhage, gastrointestinal bleeding, urinary tract hemorrhage etc. within the last 6 months
   * Surgical operation is planned that requires discontinuation of DAPT after the procedure
   * Anticoagulation therapy is underway and the risk of bleeding is high
4. Bleeding tendency due to hemorrhagic diathesis or blood coagulation disorder.
5. Left ventricular ejection fraction (LVEF) is less than 30% within 30 days before the trial registration.
6. Renal dysfunction (Creatinine value exceeds 2.0 mg/dl or in case artificial dialysis).
7. Allergy to cobalt chrome alloy or contrast agent.
8. Patients who are participating in or will planning to participate in other clinical studies that may have clinical implications for the evaluation of this trial.
9. Patients who are pregnant or breast feeding.
10. Patients who are taking Cilostazol.
11. In cases where the Investigator determines that the patient's participation in the trial is inappropriate.

<Angiographic exclusion criteria>

1. Lesion in left main coronary trunk
2. Lesion within 5 mm from the ostium right coronary artery
3. Lesion within 5 mm from the ostium left anterior descending/the ostium left circumflex branch
4. Bifurcation lesion
5. Within 1 year after implementing PCI on the target vessel or its branch
6. There are other lesions that require PCI at the time of the procedure
7. Type C of ACC / AHA classification

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-05-31 (Actual); Primary Completion 2020-03-27 (Actual); Study Completion 2024-07-26 (Actual)

PRIMARY OUTCOMES:
In-segment late lumen loss as measured by quantitative coronary angiography (QCA) | 9 months

SECONDARY OUTCOMES:
Device Success rate | Immediate post-procedure
  Device success is defined as successfully placement of the investigational stent at the target lesion, and attainment of less than 50% residual stenosis at the end of stenting.
Procedure success rate | At the time of hospital discharge, expected 1or 2 days after of procedure
  Procedure success is defined as attainment of less than 50% residual stenosis at the end of stenting and no major adverse cardiac events (death (excluding cases obviously caused by other than coronary ischemia), myocardial infarction, target lesion revascularization (TLR)) during hospitalization.
Target Lesion Failure (TLF) | 9 Months
Target Vessel Failure (TVF) | 9 Months
Stent thrombosis | 9 Months
Patient Oriented Composite End point (POCE) | 9 Months
  POCE: All cause death, all myocardial infarction, or all revascularization with ischemia
In-stent and in-segment %diameter stenosis (%DS) as measured by QCA | 9 Months
In-stent and in-segment %Angiographic Binary Restenosis (%ABR) | 9 Months
Neointima volume as measured by OCT/OFDI | 9 Months
%Volume obstruction as measured by OCT/OFDI | 9 Months
%Incomplete stent apposition (%ISA) as measured by OCT/OFDI | 9 Months
%Covered strut as measured by OCT/OFDI | 9 Months

CONTACTS AND LOCATIONS:
Locations (6):
- Japan (6):
  - Tokai University Hospital, Isehara, Kanagawa
  - Kitasato University Hospital, Sagamihara, Kanagawa
  - Saiseikai Yokohamashi Tobu Hospital, Yokohama, Kanagawa
  - Showa University Fujigaoka Hospital, Yokohama, Kanagawa
  - Mitsui Memorial Hospital, Chiyoda City, Tokyo
  - Teikyo University Hospital, tabashi City, Tokyo

IPD SHARING:
Plan to Share IPD: No